CLINICAL TRIAL: NCT04359849
Title: Sequencing and Tracking of Phylogeny in COVID-19 Study
Acronym: STOPCOVID19
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2020/34
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Investigators plan to generate a database of viral RNA sequences for SARS-CoV-2 within the Wessex region. Such whole genome data can be used to monitor mutation rates in real time and, through comparison with global databases of SARS-CoV-2 genome sequences, can be used to map transmission of the virus

DETAILED DESCRIPTION:
The current Covid-19 pandemic has caused significant strain on the health care system, and an unprecedented Governmental response to stem the spread of the disease through social distancing and self-isolation. Covid-19 is a pneumonia-like severe acute respiratory syndrome (SARS) caused by a virus, SARS-CoV-2, with similarity to the SARS virus responsible for a worldwide outbreak in 2002. Due to the original SARS outbreak, a large body of genomic data exists for SARS coronaviruses, allowing researchers to understand how the new virus SARS-CoV-2 has evolved to be so virulent in humans.

Whilst testing kits have been designed to target specific genes in the viral RNA, whole genome sequencing of the virus offers increased scope to track the epidemiology of the virus. In addition, through the use of current sequencing technology available from Oxford Nanopore Technologies (ONT), genome scanning can be performed in real time and allow for identification of specific viral variants within patient samples. As the pandemic continues to spread, understanding the evolution of the virus and its spread across the globe will help researchers to begin to predict the future spread of the virus, estimate the number of worldwide cases, and aid in the development of epidemiological models for estimating a potential end point to the pandemic crisis. In addition, the ability to track mutations in real time allows researchers access to a large body of data to explore in order to identify potential targets for cures and vaccines. These data will also feed into the design of RNA-based therapeutic targets and diagnostics using patented array technology.

In this project, the investigators aim to use Nanopore-based sequencing technology to assemble viral genomes from patients who have presented to Portsmouth Hospital NHS Trust (PHT) in the Wessex region with symptoms of Covid-19. PHT, has containment level 3 (CL3) facilities within their Microbiology Department required for inactivation of the virus and extraction of viral RNA, and has recently begun testing of potential Covid-19 patients. Viral RNA samples from patients who show positive results will be selected for sequencing using Nanopore sequencing technology. Whole genome sequences will be compared using phylogenetic analysis to identify the spread of the virus within the local area, will be analysed in the context of anonymised patient level data to look for trends in the adaptation of the virus, and will be compared with a global database of such sequences to help develop global maps of transmission.

As part of the COVID-19 Genomics UK Consortium (COG-UK), the investigators will contribute sequencing data to the consortium which will monitor changes in the virus on a national scale to understand how the virus is mutating and spreading and whether different strains are emerging

ELIGIBILITY:
Inclusion Criteria:

* Have undergone successful testing for Covid-19
* Have sufficient viral RNA remaining for research analysis following testing for Covid-19

Exclusion Criteria:

* Insufficient viral RNA remains following testing for Covid-19

Min Age: 7 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Focus on those whose tests have provided a positive result so as to maximise the number of SARS-CoV-2 genomes generated.
Sampling Method: Non-Probability Sample
Enrollment: 5602 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of whole genome sequences for the SARS-CoV-2 virus from viral RNA samples | 2 years
  Generated using Nanopore-based whole genome sequencing techniques

SECONDARY OUTCOMES:
Transmission rates of the SARS-CoV-2 virus | 2 years
  Identify mutations and viral strains prevalent within the Wessex region

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom